CLINICAL TRIAL: NCT03176654
Title: The Effect of High-Velocity Low-Amplitude Thrust Manipulation of the Cervical Spine on Pain Biomarkers in Females With Non-Specific Mechanical Neck Pain
Brief Title: The Effect of Manipulation of the Cervical Spine on Pain Biomarkers
Acronym: HVLAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Everett Lohman, D.Sc., P.T., OCS Professor Allied Health., Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 5160076
Record Dates: First submitted 2017-06-02; First posted 2017-06-05 (Actual); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Neck Pain, Posterior
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Experimental Group (HVLAT manipulation) Control Group (sham HVLAT manipulation)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVLAT manipulation (Experimental): An HVLAT manipulation is applied to the site of pain or restriction with the patient in supine. This technique uses both primary levers (pre-manipulation rotation - away (30 ° - 45 °) from the side of pain or limitation) and secondary levers (Side bending - towards coupled with lateral shift - away, and posterior-anterior (PA) shift (extension). This is a bimanual technique. For the applicator hand, the anterolateral portion of the first or second phalanx of the second ray was positioned on the superior joint partner of the target vertebrae using a cradle hold. The other hand is placed on the posterolateral aspect of the occiput (above the ear). While maintaining these positions the clinician performed the thrust with the arc of rotation dependent on the level of the target vertebrae.
  Interventions: Procedure: HVLAT manipulation
- Sham HVLAT manipulation (Sham Comparator): Subjects in the control group were instructed to lay on a table in the same position as the HVLAT manipulation group. The clinician went through the same basic steps as the HVLAT manipulation, localizing the appropriate vertebral landmarks but without carrying out the final HVLA thrust procedure.
  Interventions: Procedure: Sham HVLAT manipulation

INTERVENTIONS:
Procedure: HVLAT manipulation — HVLAT will be performed 10 minutes after the first blood draw.
  Arms: HVLAT manipulation
Procedure: Sham HVLAT manipulation — Sham HVLAT will be performed 10 minutes after the first blood draw.
  Arms: Sham HVLAT manipulation

SUMMARY:
This study evaluates the effect of high-velocity low-amplitude thrust (HVLAT) manipulation to the cervical spine on neuropeptide expression as determined by the plasma concentration of oxytocin, neurotensin, orexin A and cortisol; and Examine the effect of HVLAT manipulation on pain perception in symptomatic females with non-specific mechanical cervical spine pain

DETAILED DESCRIPTION:
A high-velocity low-amplitude thrust (HVLAT) manipulation or commonly known as a spinal manipulation, is an intervention frequently used by physical therapists and other healthcare practitioners as an alternative treatment to help relieve spinal pain The mechanism by which HVLAT manipulation modulates pain remains undefined, although this does not contradict the clinical effects from HVLAT manipulation. Furthermore, there is evidence that suggests analgesia after HVLAT manipulation. There is a variety of observed and proposed phenomena that can explain the mechanisms for the psychological, mechanical, or neurophysiological responses from a HVLAT manipulation associated with alterations in pain processing or sympathetic and motor systems' excitation.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 45 years of age
* A score of 10 or more out of 50 on the Neck Disability Index (NDI) questionnaire
* Symptoms of pain present for 30 days or less and no pain symptoms below your shoulder

Exclusion Criteria:

* Serious condition (such as cancer, spondylolisthesis, rheumatoid arthritis, or ankylosing spondylitis)
* Cervical spinal stenosis signs (such as incoordination in hands, arms and legs, inability of walking at a brisk pace, or bowel and bladder incontinence)
* Nerve root compression (such as changes in sensation, muscle weakness, or decreased reflexes)
* Works the night shift
* Steroid medication within 3 months
* Pregnancy or postpartum
* Pending legal action regarding their neck pain
* History of whiplash associated disorder and/or cervical spine surgery

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Lohman, D.Sc., Study Chair — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gross A, Miller J, D'Sylva J, Burnie SJ, Goldsmith CH, Graham N, Haines T, Bronfort G, Hoving JL; COG. Manipulation or mobilisation for neck pain: a Cochrane Review. Man Ther. 2010 Aug;15(4):315-33. doi: 10.1016/j.math.2010.04.002. Epub 2010 May 26. PMID 20510644
- [Background] Bronfort G, Haas M, Evans R, Leininger B, Triano J. Effectiveness of manual therapies: the UK evidence report. Chiropr Osteopat. 2010 Feb 25;18:3. doi: 10.1186/1746-1340-18-3. PMID 20184717

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Started | 13 | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twenty-eight female subjects with non-specific mechanical neck pain randomly assigned to one of two interventions (HVLAT or Sham HVLAT).
Groups:
- Total: Total of all reporting groups
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Customized [Mean (Full Range); unit: years] — Twenty-eight female subjects between the ages of 20 and 45 years with non-specific mechanical neck pain randomly assigned to one of two interventions (HVLAT or Sham HVLAT).
  years
    Mean age of participants | 37 [20 to 45] | 30 [20 to 45] | 37 [20 to 45]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Twenty-eight female subjects with non-specific mechanical neck pain randomly assigned to one of two interventions (HVLAT or Sham HVLAT).
  Participants | 13 | 15 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Oxytocin
Description: Samples were analyzed for Human Oxytocin, using the Multiplex Luminex-100 platform (Luminex, Inc., USA).
Time Frame: Blood will be drawn 10 minutes prior to HVLAT procedure.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Number analyzed (Participants) | 13 | 15
ug/ml | 154.5 (0.9) | 158.8 (0.5)

2. Primary Outcome: Plasma Concentration of Oxytocin
Description: Samples were analyzed for Human Oxytocin, using the Multiplex Luminex-100 platform (Luminex, Inc., USA).
Time Frame: Blood will be drawn immediately after HVLAT procedure.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Number analyzed (Participants) | 13 | 15
ug/ml | 185.1 (0.9) | 189.1 (0.5)

3. Secondary Outcome: Plasma Concentration of Neurotensin
Description: Samples were analyzed for Human Neurotensin, using the Multiplex Luminex-100 platform (Luminex, Inc., USA).
Time Frame: Within 10 minutes after consent signature completion
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Number analyzed (Participants) | 13 | 15
ug/ml | 116.0 (1.6) | 125.6 (0.2)

4. Secondary Outcome: Plasma Concentration of Neurotensin
Description: Samples were analyzed for Human Neurotensin, using the Multiplex Luminex-100 platform (Luminex, Inc., USA).
Time Frame: Blood will be drawn immediately after HVLAT procedure.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Number analyzed (Participants) | 13 | 15
ug/ml | 136.4 (1.6) | 131.6 (0.2)

5. Secondary Outcome: Plasma Concentration of Orexin A
Description: Samples were analyzed for Human Orexin A, using the Multiplex Luminex-100 platform (Luminex, Inc., USA).
Time Frame: Within 10 minutes after consent signature completion
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Number analyzed (Participants) | 13 | 15
ug/ml | 52.2 (1.0) | 62.9 (0.2)

6. Secondary Outcome: Plasma Concentration of Orexin A
Description: Samples were analyzed for Human Orexin A, using the Multiplex Luminex-100 platform (Luminex, Inc., USA).
Time Frame: Blood will be drawn immediately after HVLAT procedure.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Number analyzed (Participants) | 13 | 15
ug/ml | 73.8 (1.0) | 67.3 (0.2)

7. Secondary Outcome: Plasma Concentration of Cortisol
Description: Samples were analyzed for Human Cortisol, using the Multiplex Luminex-100 platform (Luminex, Inc., USA).
Time Frame: Within 10 minutes after consent signature completion
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Number analyzed (Participants) | 13 | 15
ug/ml | 95.8 (0.8) | 127.4 (0.5)

8. Secondary Outcome: Plasma Concentration of Cortisol
Description: Samples were analyzed for Human Cortisol, using the Multiplex Luminex-100 platform (Luminex, Inc., USA).
Time Frame: Blood will be drawn immediately after HVLAT procedure.
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
Number analyzed (Participants) | 13 | 15
ug/ml | 108.1 (0.8) | 139.7 (0.5)

ADVERSE EVENTS:
Time Frame: Subjects received a total of 1 intervention. The data collection period lasted 3 months total.
Description: The study has concluded an no subjects had any adverse events.
Arm/Group | HVLAT Manipulation | Sham HVLAT Manipulation
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

LIMITATIONS AND CAVEATS:
One limitation of this study may be the lack of a control group with no touch contact. There may be an increase in oxytocin in both groups as a consequence of the touch and pressure applied to the subject's cervical spine.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes